CLINICAL TRIAL: NCT05828901
Title: Predicting Disease Activity and Rebound Risk in MS Patients Treated With Sphingosine-1-phosphate Receptor Modulators (S1PRM)
Acronym: PATTERN
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: IM047-1034
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA tube, PAXgene tube, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Relapsing Remitting Multiple Sclerosis starting Ozanimod
  Interventions: Other: S1PR analysis on immune cells
- Relapsing Remitting Multiple Sclerosis stopping Ozanimod
  Interventions: Other: S1PR analysis on immune cells

INTERVENTIONS:
Other: S1PR analysis on immune cells — S1P receptor 1 and 5 expression will be measured on immune cells

SUMMARY:
Sphingosine 1-Phosphate (S1P) receptor modulators (S1PRMs) are part of the evolving treatment landscape of Multiple Sclerosis (MS) immunotherapies. They target the G-protein coupled S1P receptor, among other localizations expressed at the surface of lymphocytes. Binding as a functional antagonist leads to internalization of the receptor and therefore lymphocyte sequestration in the secondary lymphoid organs. The first S1PRM approved was fingolimod. More recently newer generation S1PRMs like ozanimod have been approved, which possess differences in receptor affinities, pharmacokinetics and indications (including Secondary Progressive MS or Ulcerative Colitis). Several retrospective analyses have shown that, upon cessation of fingolimod, pronounced relapse of the MS-disease called "rebound disease activity" may occur. Indeed, these relapses, sometimes with considerable severity, take place in up to 10% of patients. The risk of rebound disease of the newer generation S1PRM are not well defined.

Although of utmost importance, predictive biomarkers of treatment efficacy in general and in special circumstances, e.g. an impending rebound when S1PRM cessation is planned, are scarce.

In this prospective, exploratory observational study, we aim to investigate the predictive potential of the lymphocytic S1PR1 and 5 expression prior to treatment initiation with the newer generation S1PRM ozanimod on the future disease activity ("on treatment" part). Additionally, in a post-treatment part ("off treatment"), the incidence of rebound disease and the predictive potential of the lymphocytic S1PR1 and 5 expression will be examined in patients, where ozanimod has to be stopped due to clinical reasons.

T and B cells from patient blood samples obtained prior to treatment start/cessation and 3 - 6 months after start/cessation will be isolated and S1PR1 and 5 staining intensity will be assessed by flow cytometry (FACS). Clinical assessments (relapse assessment, EDSS, medical history etc.) will be performed at every visit and MRI evaluation, following our standard clinical and MRI MS protocol. MRI disease activity will serve as the primary endpoint for both study groups. The relationship between the flow cytometric staining intensity and the defined endpoints will be assessed statistically by using comparative statistical approaches and multivariable regression analysis where needed for both time points. The data collected will correlate the expression pattern of S1P receptors by T and B lymphocytes to the proxy of paraclinical activity as predictive biomarkers for disease activity on treatment and after treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria "On treatment":

* Adult patients with RRMS (McDonald criteria 2017) fulfilling the Swiss medic label for ozanimod
* Written informed consent

Inclusion Criteria "Off treatment":

* Adult patients with RRMS (McDonald criteria 2017) who stop ozanimod as indicated in clinical routine.
* Written informed consent

Exclusion Criteria "On treatment" and "Off treatment":

* All vulnerable persons defined by Swiss law including, but not limited to pregnant women, prisoners etc.
* Hypersensitivity and allergy against ozanimod or tablet ingredients.
* People not understanding the ICF due to mental disabilities.
* People with insufficient German or French language skills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with the diagnosis of relapsing remitting MS (RRMS), treated at the Bern University Hospital, who start or stop ozanimod treatment as indicated per clinical routine
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
"On treatment" MRI disease activity | Between 3 - 6 months after start of any new MS immunotherapy in our center compared to the previous scan
  Enhancing T1 lesions or new/enlarging T2 lesions - in the re-baseline MRI (change from baseline), defined as first MRI after treatment start performed during routine clinical care
"Off treatment" MRI disease activity | Between 3 - 6 months after start of any new MS drug in our center
  Enhancing T1 lesions or new/enlarging T2 lesions - in the re-baseline MRI of the subsequent immunotherapy after cessation of ozanimod, performed during routine clinical care

SECONDARY OUTCOMES:
"On treatment" Relapse rate | In the first year of ozanimod treatment
  Relapse rate
"Off treatment" Relapse rate and severity | In the first 6 months after ozanimod cessation
  Relapse rate (six-monthly relapse rate)
"On treatment" Disability progression | In the first year of ozanimod treatment
  Disability progression (measured as Expanded Disability Status Scale (EDSS), 9-Hole Peg Test (9-HPT), timed 25-Foot Walk Test (T25ftWT) and Symbol Digit Modalities Test (SDMT). Additional questionnaires (Fatigue Scale for Motor and Cognition (FSMC) to assess MS-related fatigue, Hospital Anxiety and Depression Scale (HADS) to assess anxiety and depression, Epworth Sleepiness Scale (ESS) to assess sleepiness and Multiple Sclerosis Impact scale (MSIS-29) to assess health-related quality of life) will be carried out.
"Off treatment" Severity | In the first 6 months after ozanimod cessation
  Severity (measured as EDSS increase during relapse) and EDSS progression in the first 6 months after ozanimod cessation will be investigated. The following exploratory endpoints will also be assessed: 9-HPT, T25ftWt, SDMT, FSMC, HADS, ESS, MSIS-29.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hoepner, PD Dr. med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Neurology department, Bern, Switzerland